CLINICAL TRIAL: NCT06302582
Title: The Efficacy and Safety of Platelet Rich Plasma Combined With Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Patients With Stage 3 and 4 Stress Injury
Brief Title: Platelet Rich Plasma Combined With Human Umbilical Cord Mesenchymal Stem Cells for Stage 3 and 4 Stress Injury
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stress injury
Record Dates: First submitted 2024-02-07; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Pressure Injuries - Stage 3; Pressure Injuries - Stage 4
Keywords: Mesenchymal stem cells; Platelet rich plasma; Pressure Injuries
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich plasma (PRP) combined with human umbilical cord mesenchymal stem cells (huMSCs) (Experimental): Inject 3ml PRP+huMSCs (5 × 106) into the edge and bottom of the wound, with 0.5 ml at each point and a distance of approximately 1-3 cm between each point. Then, apply autologous PRP gel (PRP+thrombin mixture, 2ml) evenly on the wound, with a thickness of about 2mm.
  Interventions: Biological: Platelet-rich plasma (PRP) combined with human umbilical cord mesenchymal stem cells (huMSCs)
- Control group (Other): Standard therapy
  Interventions: Other: Control group

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP) combined with human umbilical cord mesenchymal stem cells (huMSCs) — Inject 3mL PRP+huMSCs (5 × 106) into the edge and bottom of the wound, with 0.5 ml at each point and a distance of approximately 1-3 cm between each point. Then, apply autologous PRP gel (PRP+thrombin mixture, 2ml) evenly on the wound, with a thickness of about 2mm
  Arms: Platelet-rich plasma (PRP) combined with human umbilical cord mesenchymal stem cells (huMSCs)
Other: Control group — Standard therapy for patients with stage 3 and 4 stress injury
  Arms: Control group

SUMMARY:
This study is an open-label, single-center trial which aim to evaluate of efficacy and safety of human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) combined with platelet-rich plasma (PRP) in stage 3 and 4 stress injury.

DETAILED DESCRIPTION:
The 2019 edition of the International Guidelines for Clinical Prevention and Treatment of Stress Injury states that stress injury, as a globally prevalent health issue, significantly reduces the quality of life for patients and their families, increases economic burden, and leads to significant expenditure on medical resources. In recent years, the incidence and mortality rate of pressure injuries in hospitalized patients have been increasing year by year. Therefore, there is an urgent need to find a more effective treatment method for pressure injuries in clinical practice. Human umbilical cord mesenchymal stem cells (huMSCs) have immunomodulatory and anti-inflammatory effects. Platelet rich plasma (PRP) can also secrete various nutritional factors, which can effectively promote wound healing. Therefore, the combination of the two may be a more effective treatment method for pressure injuries. At present, there are few reports on the combination of PRP and huMSCs for the treatment of pressure injury. In this study, the investigators aim to evaluate the effectiveness and safety of PRP combined with huMSCs for stage 3 and 4 pressure injuries, In order to promote their clinical application.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old, regardless of gender;
* Patients with stage 3 and stage 4 pressure injuries (According to National Pressure Ulcer Advisory Panel (NPUAP)/European Pressure Ulcer Advisory Panel (EPUAP) classification system for pressure ulcers);
* There were no complications affecting the wound healing;
* After through debridement for the first time, the wound volume meets the requirement of "10-100cm3"; Platelet count before treatment 100~300×109/L;
* The patient voluntarily participates and signs an informed consent form.

Exclusion Criteria:

* Individuals with coagulation dysfunction or hemorrhagic diseases;
* People with skin diseases, diabetes and immune diseases;
* Individuals with mental or psychological disorders;
* Individuals with allergies to multiple drugs;
* Pregnant or lactating women;
* Those who need to take medication that affects platelet and coagulation function for a long time or in the near future, but have not stopped taking medication within the past week.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pressure Ulcer Scale for Healing (PUSH) | Baseline,1,2,4 and 6 weeks
  The scale includes three dimensions: wound area, exudate volume, and tissue type. The total score of the three dimensions was indicated the healing of pressure injury and ranged from 0 to 17 points, with 0 points indicating wound healing. The PUSH score decreased, indicating improvement. The total score increased, indicating deterioration. Multiple pressure injuries in the same patient were evaluated separately.
Change from baseline in Determination of growth factor content | Baseline,1, 2 and 3 weeks
  Serum epidermal growth factor (EGF) and vascular endothelial growth factor (VEGF) were detected during treatment.

SECONDARY OUTCOMES:
Wound healing time | up to 4 months
  The wound healing standard is wound closure and epithelial tissue coverage, and the wound healing time refers to the time from the date of direct treatment to wound healing for the patient. The wound healing time was recorded through dressing change in outpatient department or phone call follow-up.
Positive rate of bacterial culture | Baseline and 2 weeks
  The patient's wound secretions were collected for bacterial culture on the day of stem cell treatment and 2 weeks after treatment.

OTHER OUTCOMES:
Safety evaluation | up to 1 week
  Any adverse events that occur during the treatment process must be recorded in detail. The record of adverse events should include a description of the adverse event and all related symptoms, the time of occurrence, severity, duration, measures taken, and the final outcome and outcome, as well as an evaluation of the possible correlation between the adverse event and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Central laboratory, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daneste H, Mohammadzadeh Boukani L, Ramezani N, Asadi F, Zaidan HK, Sadeghzade A, Ehsannia M, Azarashk A, Gholizadeh N. Combination therapy along with mesenchymal stem cells in wound healing; the state of the art. Adv Med Sci. 2023 Sep;68(2):441-449. doi: 10.1016/j.advms.2023.10.006. Epub 2023 Nov 2. PMID 37924749
- [Result] Qu S, Hu Z, Zhang Y, Wang P, Li S, Huang S, Dong Y, Xu H, Rong Y, Zhu W, Tang B, Zhu J. Clinical Studies on Platelet-Rich Plasma Therapy for Chronic Cutaneous Ulcers: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Adv Wound Care (New Rochelle). 2022 Feb;11(2):56-69. doi: 10.1089/wound.2020.1186. Epub 2021 Jun 8. PMID 33607926
- [Result] Kunder V, Sharma KC, Rizvi Z, Soubelet R, Ducharme M. The Use of Platelet-Rich Plasma in the Treatment of Diabetic Foot Ulcers: A Scoping Review. Cureus. 2023 Aug 14;15(8):e43452. doi: 10.7759/cureus.43452. eCollection 2023 Aug. PMID 37711926
- [Result] Rainys D, Cepas A, Dambrauskaite K, Nedzelskiene I, Rimdeika R. Effectiveness of autologous platelet-rich plasma gel in the treatment of hard-to-heal leg ulcers: a randomised control trial. J Wound Care. 2019 Oct 2;28(10):658-667. doi: 10.12968/jowc.2019.28.10.658. PMID 31600109
- [Result] Wang Y, Luan S, Yuan Z, Wang S, Fan S, Ma C, Wu S. The Combined Use of Platelet-Rich Plasma Clot Releasate and Allogeneic Human Umbilical Cord Mesenchymal Stem Cells Rescue Glucocorticoid-Induced Osteonecrosis of the Femoral Head. Stem Cells Int. 2022 May 2;2022:7432665. doi: 10.1155/2022/7432665. eCollection 2022. PMID 35547633